CLINICAL TRIAL: NCT07093216
Title: Understanding Response Variability to Optimize Exercise Efficacy for Improving Health Among Older Adults
Brief Title: Healthy Aging Through Optimized Exercise
Acronym: HELIOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Thomas W. Buford, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 300013021
Record Dates: First submitted 2025-07-14; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Aging
Keywords: Intrinsic Capacity; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose (Experimental): Testing Dose of Exercise
  Interventions: Behavioral: Exercise
- Intensity (Experimental): Testing Intensity of Effort
  Interventions: Behavioral: Exercise
- Mode (Experimental): Resistance vs Aerobic
  Interventions: Behavioral: Exercise
- Volume (Experimental): Amount of Exercise Performed
  Interventions: Behavioral: Exercise
- Time of Day (Experimental): Time of Day Exercise Performed
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 6 month exercise intervention

SUMMARY:
here is enormous variation in how individuals respond to exercise and understanding the factors that drive this variation will guide individualized exercise prescriptions to improve or maintain health into older age. This study will help to elucidate reasons for the variation in the responses to exercise in older adults.

DETAILED DESCRIPTION:
here is enormous variation in how individuals respond to exercise and understanding the factors that drive this variation will guide individualized exercise prescriptions to improve or maintain health into older age. Our multidisciplinary team will apply Multiphase Optimization Strategy Framework (MOST) principles to addresses the impacts of exercise intervention components (e.g. exercise timing, aerobic exercise intensity levels, resistance exercise intensity levels, and training volume levels), as well as participant-specific factors (e.g. age, sex, race, BMI, and medication use), on health domains of Intrinsic Capacity (locomotion, vitality, sensory, psychological, and cognition) among older adults in response to six months of supervised, center-based exercise training. This approach - unprecedented in the fields of exercise and aging - will provide comprehensive evidence to more fully understand the variation in the responses to exercise in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study procedure
* 60+ years of age
* <120 min/wk of self-reported moderate physical activity as assessed by Community Health Activities Model Program for Seniors (CHAMPS) physical activity questionnaire13
* Evidence of impairment in one or more Intrinsic Capacity domains (see section 3.2)
* Passage of a physical exam and diagnostic, graded exercise test with 12-lead ECG reviewed by a cardiologist or otherwise credentialed clinician.

Exclusion Criteria:

* End-stage disease and/or a life expectancy less than one year
* Resistant hypertension, defined as BP > 140/90, despite the use of three or more anti-hypertensive drugs
* Chronic kidney disease
* Serum creatinine >2.5 mg/dL in men or >2.0 mg/dL in women
* Serum potassium >5.0 mEq/L
* Urinary protein > 1 on dipstick
* Abnormal liver enzymes (AST, ALT, or alkaline phosphatase > 2.5 times the upper limit of normal)
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Acute myocardial infarction identified by ECG
* Current treatment for malignancy
* Known diagnosis of dementia
* Any other disease or condition that would preclude completion of all testing and exercise training
* Any other condition that would interfere with testing or increase risk of complications during exercise
* Any other condition or events considered exclusionary by the PIs and/or study clinicians.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2031-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Intrinsic Capacity | 6 months
  Single composite score of results of multiple tests across five domains: 1) Locomotion, 2) Vitality, 3) Sensory, 4) Psychological, and 5) Cognition

IPD SHARING:
Plan to Share IPD: Undecided